CLINICAL TRIAL: NCT04150367
Title: Open-label, Randomized, Multicenter, Controlled, Parallel, Comparative Study of Efficacy and Safety of Treatment of Tuberculosis With Isoniazid, Rifampicin, Ethambutol for Intravenous Infusion in Comparison With Oral Forms While the Intensive Phase of Treatment for Patients With Widespread Destructive Pulmonary Tuberculosis With Bacterial Excretion.
Brief Title: Efficacy and Safety of Intravenous Treatment of Tuberculosis
Status: Terminated | Type: Observational
Why Stopped: According to Sponsor decision.
Sponsor: Yuria-Pharm (Industry)
Responsible Party: Sponsor
Other Study IDs: Invent-1
Record Dates: First submitted 2017-10-25; First posted 2019-11-04 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Isoniazid; Rifampin; Solutions; Ethambutol; Tablets

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with first diagnosed widespread destructive pulmonary tuberculosis with bacterial excretion, who receive intravenous treatment with Isoniazid, Rifampicin, Ethambutol first two months of intensive phase of tuberculosis treatment. Then group receives oral treatment of tuberculosis according to the known scheme.
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Ethambutol
- Control group: Patients with first diagnosed widespread destructive pulmonary tuberculosis with bacterial excretion, who receive oral forms of Isoniazid, Rifampicin, Ethambutol first two months of intensive phase of tuberculosis treatment. Then group receives oral treatment of tuberculosis according to the known scheme.
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Ethambutol

INTERVENTIONS:
Drug: Isoniazid — Solution for injections, 100 mg/ml, 5 ml. Participants will get the dosage according to the instruction for use.
  Other Names: Bitub
  Groups: Study group
Drug: Rifampicin — Participants will get the dosage according to the instruction for use.
  Other Names: Rifampin, Lyophilisate for solution for infusion 600 mg.
  Groups: Study group
Drug: Ethambutol — Participants will get the dosage according to the instruction for use.
  Other Names: Inbutol, Solution for injections100 mg/ml, 20 ml.
  Groups: Study group
Drug: Rifampicin — Participants will get the dosage according to the instruction for use.
  Other Names: Rifampicin 150 mg Capsules
  Groups: Control group
Drug: Isoniazid — . Participants will get the dosage according to the instruction for use.
  Other Names: Isoniazid, Tablets, 300mg.
  Groups: Control group
Drug: Ethambutol — Participants will get the dosage according to the instruction for use.
  Other Names: Ethambutol, Tablets 400 mg.
  Groups: Control group

SUMMARY:
This Open-label, Randomized, Multicenter, Controlled, Parallel, Comparative Study will compare the efficacy and safety of intravenous treatment with Isoniazid, Rifampicin, Ethambutol first two months of intensive phase of tuberculosis treatment and the treatment with the oral forms of Isoniazid, Rifampicin, Ethambutol first two months of intensive phase of tuberculosis treatment for Patients With Widespread Destructive Pulmonary Tuberculosis With Bacterial Excretion.

DETAILED DESCRIPTION:
There are two groups of patients with first diagnosed widespread destructive pulmonary tuberculosis with bacterial excretion. The first group receives intravenous treatment with Isoniazid, Rifampicin, Ethambutol first two months of intensive phase of tuberculosis treatment. The second group gets oral forms of Isoniazid, Rifampicin, Ethambutol first two months of intensive phase of Tuberculosis treatment. Then both groups receive oral treatment of tuberculosis according to the known scheme.

Up to 318 participants will be randomized into this study, with 159 participants being randomized to the control arm and 159 participants being randomized to the experimental arm. It Supposed that not less than 254 participants will finish the study (about 127 participants in each arm) and their results will be included in the statistical analysis.

While the intensive phase participants of both arms will be hospitalized in the Tuberculosis Dispensary.

ELIGIBILITY:
Inclusion Criteria:

1. men and women;
2. The age of 18 - 65 years inclusive;
3. Patients diagnosed with: first diagnosed pulmonary tuberculosis;
4. Patients with at least one positive result of a microbiological study of the sputum on the Mycobacterium tuberculosis (during the screening, the results of a microbiological sputum examination on an Mycobacterium tuberculosis up to 7 days old can be used);
5. Patients with radiographically and optionally CT confirmed cavity / cavities of destruction in the lungs, as well as a widespread tuberculosis process (occupying at least 2 segments of the lungs) (during the screening, the results of X-ray examination of the chest up to 7 days old can be used );
6. For women with reproductive potential - negative result of urine test for pregnancy and consent to use a reliable method of contraception before the end of the study;
7. Provided informed written consent of the patient to participate in the study;
8. The patient's ability to adequately cooperate in the research process;
9. Patients with negative analysis of GenXpert MBT / RIF (at the time of screening, analysis results not older than 7 days may be used);
10. Oral consent of the patient to stop using alcohol during the study period.

Exclusion Criteria:

1. Patients who, according to the results of a sputum test using the GenXpert MBT / RIF method, are determined to be resistant to rifampicin.
2. Pregnancy, lactation;
3. Epilepsy and other diseases, which are accompanied by a tendency to convulsive seizures;
4. Severe psychosis;
5. Poliomyelitis (including in the anamnesis);
6. Diseases of the cardiovascular system, respiratory system, diabetes mellitus, impaired liver function, kidney, thyroid gland, vision, the presence of concomitant diseases or acute conditions, which, according to the researcher, do not allow the patient to participate in this study;
7. HIV infection;
8. Intolerance (including history) of any of the drugs studied;
9. Participation in any other clinical trial at the time of inclusion in this study and for the last 30 days before the date of screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with first diagnosed widespread destructive pulmonary tuberculosis with bacterial excretion.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-07-14 (Actual); Study Completion 2018-07-14 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with negative results of sputum analysis on Mycobacterium tuberculosis . | Тhe end of the 1st month from the start of treatment (after taking 30 doses of each drug by the patient)
  Percentage of patients with negative results of sputum analysis on Mycobacterium tuberculosis in the main and control groups.

SECONDARY OUTCOMES:
Time until the negative result of the Mycobacterium tuberculosis tests is obtained. | 2 weeks - 3 months
  Time until the negative result of sputum Mycobacterium tuberculosis tests is obtained for each patient.
Combined percentage ratio of patients with negative results of Mycobacterium tuberculosis analysis and clinical improvement. | 2 months after the start of treatment (after taking the patient 60 doses of each preparation of the intensive phase).
  Combined percentage ratio of patients who have negative results of sputum analysis on Mycobacterium tuberculosis and clinical improvement at the same time.
Combined percentage of patients with no response to treatment in 12 months. | 12 months after the start of treatment (13 months after initiation of treatment for patients who still have the positive results of the sputum analysis on Mycobacterium tuberculosis after taking 60 doses of each preparation of the intensive phase).
  Combined percentage ratio of patients with no response to treatment in 12 months.
Combined percentage ratio of patients with no response to treatment in 18 months. | 18 months after the start of treatment (19 months after initiation of treatment for patients who still have the positive results of the sputum analysis on Mycobacterium tuberculosis after taking 60 doses of each preparation of the intensive phase).
  Combined percentage ratio of patients with no response to treatment in 18 months.
Combined percentage ratio of patients with relapse of active tuberculosis in 18 months. | 18 months after the start of treatment (19 months after initiation of treatment for patients who still have the positive results of the sputum analysis on Mycobacterium tuberculosis after taking 60 doses of each preparation of the intensive phase).
  Combined percentage ratio of patients with relapse of active tuberculosis in 18 months.
Combined percentage ratio of patients with death due to active tuberculosis in 18 months. | 18 months after the start of treatment (19 months after initiation of treatment for patients who still have the positive results of the sputum analysis on Mycobacterium tuberculosis after taking 60 doses of each preparation of the intensive phase).
  Combined percentage ratio of patients with death due to active tuberculosis in 18 months.
Combined percentage ratio of patients with relapse of active tuberculosis in 12 months. | 12 months after the start of treatment (13 months after initiation of treatment for patients who still have the positive results of the sputum analysis on Mycobacterium tuberculosis after taking 60 doses of each preparation of the intensive phase).
  Combined percentage ratio of patients with relapse of active tuberculosis in 12 months.
Combined percentage ratio of patients with death due to active tuberculosis in 12 months. | 12 months after the start of treatment (13 months after initiation of treatment for patients who still have the positive results of the sputum analysis on Mycobacterium tuberculosis after taking 60 doses of each preparation of the intensive phase).
  Combined percentage ratio of patients with death due to active tuberculosis in 12 months.

OTHER OUTCOMES:
Percentage ratio of severe adverse events. | From 1 week till 7 months after the start of treatment.
  All kinds of adverse events.
Comparative cost of treatment of the main disease and complications at 6 months after the start of the treatment. | 6 months after the start of treatment/
  Comparative cost of treatment of the main disease and complications based on the average cost of all medical services for the medical institutions participating in the study at 6 months after the start of treatment.
Comparative cost of treatment of the main disease and complications at 12 months after the start of the treatment. | 12 months after the start of treatment
  Comparative cost of treatment of the main disease and complications based on the average cost of all medical services for the medical institutions participating in the study at 12 months after the start of treatment.
Comparative cost of treatment of the main disease and complications at 18 months after the start of the treatment. | 18 months after the start of treatment
  Comparative cost of treatment of the main disease and complications based on the average cost of all medical services for the medical institutions participating in the study at 18 months after the start of treatment.

CONTACTS AND LOCATIONS:
Locations (9):
- Ukraine (9):
  - Regional Clinical Antituberculosis Dispensary, Chernivtsi
  - Regional phthisiopulmonary center, Ivano-Frankivsk
  - Regional Antituberculosis Dispensary №1, Kharkiv
  - Regional Antituberculosis Dispensary, Kherson
  - National Yanovsky's Institute of Phthisiology and Pulmonology, Kyiv
  - Regional territorial medical anti-tuberculosis association, Lutsk
  - Lviv Regional Phthisiopneumological Clinical Treatment and Diagnostic Center, Lviv
  - Regional Clinical Antituberculosis Dispensary, Sumy
  - Ternopil Regional TB Dispensary, Ternopil

IPD SHARING:
Plan to Share IPD: Undecided